CLINICAL TRIAL: NCT03474042
Title: A Phase IIa, Randomized, Double-blind, Placebo-controlled Study to Evaluate GLPG2737 in Orkambi-treated Subjects With Cystic Fibrosis Homozygous for the F508del Mutation
Brief Title: GLPG2737 on Top of Orkambi in Subjects With Cystic Fibrosis
Acronym: PELICAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG2737-CL-202; 2017-002181-42 (EudraCT Number)
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLPG2737 (Experimental): GLPG2737 will be provided as capsules for oral use.
  Interventions: Drug: GLPG2737
- Placebo (Placebo Comparator): Placebo will be provided as capsules for oral use.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG2737 — GLPG2737 oral capsules administered twice daily for 28 days on top of Orkambi.
  Arms: GLPG2737
Drug: Placebo — Placebo oral capsules administered twice daily for 28 days on top of Orkambi.
  Arms: Placebo

SUMMARY:
This is a Phase IIa, multi-center, randomized, double-blind, placebo-controlled, parallel-group study to evaluate GLPG2737 administered orally b.i.d. for 28 days to adult male and female subjects with a confirmed diagnosis of cystic fibrosis homozygous for the F508del CFTR mutation and on stable treatment with Orkambi.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject ≥18 years of age on the day of signing the ICF.
* A confirmed clinical diagnosis of CF and homozygous for the F508del CFTR mutation.
* Stable intake of physician prescribed Orkambi (lumacaftor 400 mg/ivacaftor 250 mg b.i.d.) for at least 12 weeks prior to the first study drug administration, and planned continuation of Orkambi for the duration of the study.
* FEV1 ≥40% of predicted normal for age, gender and height at screening (pre- or postbronchodilator).
* Sweat chloride concentration ≥60 mmol/L at screening.

Exclusion Criteria:

* History of serious allergic reaction to any drug as determined by the investigator (e.g., anaphylaxis requiring hospitalization) and/or known sensitivity to any component of the study drug.
* History of clinically meaningful unstable or uncontrolled chronic disease that makes the subject unsuitable for inclusion in the study in the opinion of the investigator.
* Unstable pulmonary status or respiratory tract infection (including rhinosinusitis) requiring a change in therapy within 4 weeks prior to the first study drug administration.
* History of hepatic cirrhosis with portal hypertension (e.g.,signs/symptoms of splenomegaly, esophageal varices, etc.).
* Abnormal liver function test at screening, defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) and/or alkaline phosphatase and/or gammaglutamyl transferase (GGT) ≥3 x the upper limit of normal (ULN), and/or total bilirubin ≥1.5 x the ULN at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sweat chloride concentration compared to placebo | Between day 1 pre-morning dose and Day 28.
  To assess Change from baseline in sweat chloride concentration compared to placebo.

SECONDARY OUTCOMES:
Change versus placebo in the proportion of subjects with adverse events. | Between Day 1 and 3 weeks after the last dose.
  To assess safety and tolerability by the number and percentage of subjects with adverse events.
Change from baseline in sweat chloride concentration. | From baseline (pre-morning dose on Day 1) through 28 days.
  To assess the change from baseline in sweat chloride concentration.
Change in percent predicted forced expiratory volume in 1 second (FEV1). | From baseline (pre-morning dose on Day 1) through 28 days.
  To assess the change from baseline in percent predicted forced expiratory volume in 1 second (FEV1).
Change in the respiratory domain of the cystic fibrosis questionnaire-revised (CFQ-R). | From baseline (pre-morning dose on Day 1) through 28 days.
  To assess the change from baseline in the respiratory domain of the cystic fibrosis questionnaire-revised (CFQ-R).
Maximum observed plasma concentration of GLPG2737 (Cmax) | Between day 1 pre-dose and day 14.
  To characterize the PK of GLPG2737 and its active metabolite, ivacaftor, and lumacaftor.
Area under the plasma concentration-time curve from time zero until 8 hours (AUC0-8h) post-dose calculated by the linear up - logarithmic down trapezoidal rule (on Day 14) | Between day 1 pre-dose and day 14.
  To characterize the PK of GLPG2737 and its active metabolite G1125498 (M4), ivacaftor, and lumacaftor.
Trough plasma concentration observed at the end of the dosing interval (Ctrough). | Between day 1 pre-dose and day 28.
  To characterize the PK of GLPG2737 and its active metabolite G1125498 (M4), ivacaftor, and lumacaftor.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Van de Steen, MD MBA, Study Director — Galapagos NV
Locations (9):
- Germany (9):
  - Study Site II, Berlin
  - Study Site V, Cologne
  - Study Site X, Dresden
  - Study Site III, Essen
  - Study Site IV, Frankfurt
  - Study Site I, Heidelberg
  - Study Site VI, München
  - Study Site IX, Stuttgart
  - Study Site VIII, Tübingen

REFERENCES:
- [Derived] van Koningsbruggen-Rietschel S, Conrath K, Fischer R, Sutharsan S, Kempa A, Gleiber W, Schwarz C, Hector A, Van Osselaer N, Pano A, Corveleyn S, Bwirire D, Santermans E, Muller K, Bellaire S, Van de Steen O. GLPG2737 in lumacaftor/ivacaftor-treated CF subjects homozygous for the F508del mutation: A randomized phase 2A trial (PELICAN). J Cyst Fibros. 2020 Mar;19(2):292-298. doi: 10.1016/j.jcf.2019.09.006. Epub 2019 Oct 5. PMID 31594690